CLINICAL TRIAL: NCT02059889
Title: Diffusion-weighted MRI for Individualized Radiation Therapy Planning of Lung Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: slow accrual
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MCC-13-09531; HM20000190 (Other: VCU IRB); MCC20000190 (Other: VCU Massey Cancer Center); NCI-2014-00113 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2014-02-07; First posted 2014-02-11 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Recurrent Non-small Cell Lung Cancer; Stage IIA Non-small Cell Lung Cancer; Stage IIB Non-small Cell Lung Cancer; Stage IIIA Non-small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer
Keywords: Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Diffusion Magnetic Resonance Imaging; Four-Dimensional Computed Tomography; Fluorodeoxyglucose F18; Positron-Emission Tomography; Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic (diffusion-weighted MRI, 4D CT, FDG-PET) (Experimental): Patients undergo 15 imaging studies: 5 chest CT scans, 5 chest MRI scans, 5 PET scans. Each scan will be obtained before treatment begins, weeks 2 and 4 during radiation therapy, 3 months and 1 year following radiation therapy. THe chest CT obtained pre-treatment, at 3 months post treatment and 1 year post treatment are considered routine and would be obtained regardless of study participation. The pre-treatment PET scan is also considered routine. All other scans are being done for the purposes of this research.
  Interventions: Device: diffusion-weighted magnetic resonance imaging; Device: 4-dimensional computed tomography; Radiation: fludeoxyglucose F 18; Device: FDG-PET

INTERVENTIONS:
Device: diffusion-weighted magnetic resonance imaging — Undergo diffusion-weighted MRI
  Other Names: diffusion-weighted MRI
Device: 4-dimensional computed tomography — Undergo 4D CT
  Other Names: 4D-CT
Radiation: fludeoxyglucose F 18 — Undergo FDG-PET
  Other Names: 18FDG, 2-F18-fluoro-2-deoxyglucose, 63503-12-8, FDG, Fluorine-18 2-Fluoro-2-deoxy-D-Glucose, fluorodeoxyglucose F 18, Fluorodeoxyglucose F18
Device: FDG-PET — Undergo FDG-PET
  Other Names: FDG-PET, PET, PET scan, tomography, emission computed

SUMMARY:
This clinical trial studies diffusion-weighted magnetic resonance imaging (MRI) in identifying and localizing tumors in patients with non-small cell lung cancer undergoing radiation therapy. Diagnostic procedures such as diffusion weighted MRI may help identify where active cancer is to improve the targeting accuracy of radiotherapy. Comparing results of diagnostic procedures done before, during, and after radiation therapy may help determine how the location and volume of tumors changes over time and predict how the tumor will respond to therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess diffusion-weighted MRI as an early predictor for tumor response in patients with non-small cell lung cancer (NSCLC).

II. Establish the potential of individualized radiotherapy targeting of radioresistant tumor sub-volumes.

OUTLINE:

Patients undergo diffusion-weighted MRI within 4 weeks of radiation start (baseline), during the second week of radiation therapy, during the fourth week of radiation therapy, and at 3 months after radiation therapy (post-treatment). Patients also undergo standard of care 4-dimensional (4D) computed tomography (CT) and fludeoxyglucose F 18 (FDG)-positron emission tomography (PET) at the same time points.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be able to undergo MRI imaging; contrast application will be determined according to institutional guidelines; patients with lung cancer or locally recurrent lung cancer (following surgery) who are scheduled to receive external beam radiation therapy for at least 6 weeks
* Tumor visible on planning CT scan
* Negative pregnancy test for women of childbearing potential prior to study entry

Exclusion Criteria:

* Patients requiring continuous supplemental oxygen
* Patients with metal implants including pace makers and defibrillators
* Patients with cerebral aneurysm clips or middle ear implant
* Patients with pain pump, a programmable shunt, or non-surgical metal (i.e. a foreign body)
* Claustrophobic patients
* Prior radiotherapy to body area under investigation
* No vulnerable populations will be enrolled (prisoners, children, pregnant females, or institutionalized individuals)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Measurement of gross tumor volume and involved lymph nodes | Up to 3 months
  A paired sample t-test could be applied to test the difference between MRI, CT, and PET-CT contours. Parameters used for comparison will include volume size, volume overlap, such as Dice similarity coefficients and Jaccard index, and surface distance maps including Hausdorff distance.
Change in functional response | Baseline to 3 months
  Patients will be classified into responders and non-responders based on their PET signal which will serve as the reference method for response assessment. Although this is a little different from the three group analysis of variance (ANOVA) used in the power calculation, it is expected that there will be similar high power when the partial responders and non-responders are combined. Receiver operating characteristic (ROC) analysis will be used to define a threshold of apparent diffusion coefficient (ADC) change to stratify between metabolic responders vs. non-responders.
Spatial concordance of multimodality imaging for whole image registration | Up to 3 months
  A paired sample t-test will be used.
Temporospatial registrations of radioresistant sub-volumes | Up to 3 months
  A paired sample t-test will be used. ROC analysis will be performed only for radioresistant sub-volumes to identify which diffusion weighted-MRI functional signal thresholds correlate with levels of tumor activity defined on PET.

SECONDARY OUTCOMES:
Change in ADC | Baseline to 4 weeks
  Fourth week ADC change will be compared to metabolic response defined by the fourth week PET using three group ANOVA and ROC analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Weiss, MD, Principal Investigator — Massey Cancer Center
Locations (1):
- Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia, United States